CLINICAL TRIAL: NCT01497834
Title: A Phase 3 Japanese Study of BMS-790052 Plus BMS-650032 Combination Therapy in Chronic Hepatitis C Genotype 1b Infected Subjects Who Are Non Response to Interferon Plus Ribavirin and Interferon Based Therapy Ineligible Naive/Intolerant
Brief Title: A Phase 3 Study in Combination With BMS-790052 and BMS-650032 in Japanese Hepatitis C Virus (HCV) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI447-026
Record Dates: First submitted 2011-12-02; First posted 2011-12-23 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daclatasvir + Asunaprevir (Experimental)
  Interventions: Drug: BMS-790052 (Daclatasvir); Drug: BMS-650032 (Asunaprevir)

INTERVENTIONS:
Drug: BMS-790052 (Daclatasvir) — Tablets, Oral, 60mg, Once daily, 24 weeks
Drug: BMS-650032 (Asunaprevir) — Capsules, Oral, 100mg, Twice daily, 24 weeks

SUMMARY:
The purpose of this study is to assess the anti-viral activity of BMS-790052 and BMS-650032 combination therapy in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-1b infected patient
* HCV RNA viral load of ≥ 100,000 IU/mL at screening
* Ages 20 to 75 years
* Non-responder to Interferon plus Ribavirin therapy
* Patient who has been excluded from interferon/ribavirin therapy or intolerant for Interferon/Ribavirin therapy

Exclusion Criteria:

Patients who have -

* Hepatocellular carcinoma
* Co-infection with Hepatitis B virus (HBV) or Human Immunodeficiency Virus (HIV)
* Severe or uncontrollable complication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Antiviral activity, as determined by the proportion of subjects with SVR24 | After 24 weeks of the last dose
  SVR24 - sustained virologic response at follow-up Week 24 (after end of treatment)

SECONDARY OUTCOMES:
Antiviral activity, as determined by the proportion of subjects who achieve Hepatitis C virus (HCV) ribonucleic acid (RNA) below lower limit of quantitation (LLOQ) target detected or not detected | Weeks 1, 2, 4, 6, 8, 10 and 12; Weeks 4 and 12; End of treatment (EOT), or post treatment Week 12
Antiviral activity, as determined by the proportion of subjects who achieve HCV RNA below LLOQ, target not detected | Weeks 1, 2, 4, 6, 8, 10 and 12; Weeks 4 and 12; EOT, or post treatment Week 12, post treatment Week 24
Safety, as measured by the frequency of serious adverse events (SAEs), discontinuations due to adverse events (AEs), AEs by intensity and laboratory abnormalities by toxicity grade | End of treatment plus 7 days
Proportion of subjects with SVR24 by IL28B status [CC, CT, or TT genotype at the IL28B rs12979860 single nucleotide polymorphisms (SNP)] | Follow-up Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- Japan (24):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Amagasaki-shi, Hyōgo
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kawasaki-Shi, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Suita, Osaka
  - Local Institution, Suita-shi, Osaka
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Shinagawa-ku, Tokyo
  - Local Institution, Chuo-shi, Yamanashi

REFERENCES:
- [Derived] Hernandez D, Yu F, Huang X, Kirov S, Pant S, McPhee F. Impact of Pre-existing NS5A-L31 or -Y93H Minor Variants on Response Rates in Patients Infected with HCV Genotype-1b Treated with Daclatasvir/Asunaprevir. Adv Ther. 2016 Jul;33(7):1169-79. doi: 10.1007/s12325-016-0354-1. Epub 2016 Jun 10. PMID 27287851
- [Derived] Kao JH, Jensen DM, Manns MP, Jacobson I, Kumada H, Toyota J, Heo J, Yoffe B, Sievert W, Bessone F, Peng CY, Roberts SK, Lee YJ, Bhore R, Mendez P, Hughes E, Noviello S. Daclatasvir plus asunaprevir for HCV genotype 1b infection in patients with or without compensated cirrhosis: a pooled analysis. Liver Int. 2016 Jul;36(7):954-62. doi: 10.1111/liv.13049. Epub 2016 Jan 24. PMID 26683763
- [Derived] Kumada H, Suzuki Y, Ikeda K, Toyota J, Karino Y, Chayama K, Kawakami Y, Ido A, Yamamoto K, Takaguchi K, Izumi N, Koike K, Takehara T, Kawada N, Sata M, Miyagoshi H, Eley T, McPhee F, Damokosh A, Ishikawa H, Hughes E. Daclatasvir plus asunaprevir for chronic HCV genotype 1b infection. Hepatology. 2014 Jun;59(6):2083-91. doi: 10.1002/hep.27113. Epub 2014 Apr 1. PMID 24604476
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx